CLINICAL TRIAL: NCT04871815
Title: Preliminary Examination of the Effects of Sodium Pyruvate Nasal Spray (N115) on Symptoms Associated With COVID19 Long Haulers.
Brief Title: Effects of Sodium Pyruvate Nasal Spray in COVID-19 Long Haulers.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cellular Sciences, inc. (Industry)
Collaborators: Missouri State University (Other); Dynamic DNA Laboratories (Industry); Trinity Health System (Industry); Family First Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI-COVID-19_009
Record Dates: First submitted 2021-04-27; First posted 2021-05-04 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Long COVID
Keywords: COVID19, Long Haulers
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: All subjects will be monitored for 1 week without intervention to obtain a baseline for signs and symptoms associated with COVID19 Long Haulers. All subjects will then be monitored for an additional week for signs and symptoms of COVID19 Long Haulers while using the N115 sodium pyruvate nasal spray 3x daily for that week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment of COVID19 Long Haulers with sodium pyruvate nasal spray (Experimental): This is a single arm, open label study. All subjects will be provided a log for monitoring symptoms associated with Long COVID and asked to record symptom severity using a likert scale for one week. All subjects will then use N115 sodium pyruvate nasal spray 3x daily for an additional week and continue to log their symptoms.
  Interventions: Drug: sodium pyruvate nasal spray

INTERVENTIONS:
Drug: sodium pyruvate nasal spray — Subjects will use a sodium pyruvate nasal spray 3x daily for 7 days.
  Other Names: N115

SUMMARY:
There are approximately 12 million Americans with COVID-19 Long Hauler Symptoms, including athletes. The symptoms include hypoxemia (low SaO2), fatigue, coughing/sneezing, dyspnea, trouble breathing, body aches, headaches. This chronic disease is referred to as COVID-19 Long Haulers. 7-10% of COVID-19 long haulers are also at serious risk of developing Pulmonary Fibrosis. Conversely, patients with Pulmonary Fibrosis have an increased risk and susceptibility to COVID-19 infection, which can reach a mortality rate of 50%. In a Phase III Clinical Trial in patients in Pulmonary Fibrosis and Idiopathic pulmonary fibrosis, the inhalation of the sodium pyruvate nasal spray demonstrated a statistically and clinically significant improvement in all lung functions, compared to baseline, including an increase in FEV-1, SaO2, FVC, FEV-1/FVC ratios (from 52% to 86%) and a reduction in coughing and fatigue. EmphyCorp/Cellular Sciences Inc. has submitted over 17 human clinicals (Phase I, II, III including animal safety data) to the FDA, demonstrating that the inhalation of sodium pyruvate, significantly reduced respiratory and nasal Inflammation, including oxygen radicals and inflammatory cytokines including IL-6, that causes the so-called cytokine storm COVID-19 patients. Thousands of patients treated with inhaled sodium pyruvate including patients with COPD, Pulmonary Fibrosis, CF, Allergic Rhinitis, Chronic Rhinitis, Sinusitis, and Flu, demonstrated statistically and clinically significant improvement in lung functions with no adverse events reported. This study will examine the effects of N115 (Sodium pyruvate nasal spray) treatment on the symptoms associated with COVID-19 Long Haulers.

DETAILED DESCRIPTION:
In numerous human clinical trials (17, phase I, II, III clinical trials) submitted to the FDA, for COPD, Pulmonary Fibrosis, CF, Allergic Rhinitis, Chronic Rhinitis, Sinusitis, and Flu patients, inhaled sodium pyruvate reduced nasal and lung inflammation and congestion by reducing inflammatory cytokines including the IL-6 cytokine that causes the so-called cytokine storm with no known adverse reactions. Cellular Sciences received Orphan Drug Designations for Pulmonary Fibrosis and Cystic Fibrosis. Mice studies conducted by Dr. Lupfer at Missouri State University substantiated our finding by testing nebulized sodium pyruvate in flu (influenza A H1N1 virus) infected mice that decreased morbidity, weight loss, proinflammatory cytokines, and decreased viral titers (virus numbers) compared to the Saline Placebo Control. Additionally, treated mice consumed more chow during infection indicating improved symptoms (same results reported in a pilot mice COVID-19 study). There were notable improvements in pro-inflammatory cytokine production (IL-1β) and lower virus titers (viral numbers) on days 7 post infection in mice treated with Sodium pyruvate compared to the Saline Placebo Control animals. As pyruvate acts on the host immune response, metabolic pathways and not directly on the virus, our data demonstrate that sodium pyruvate is a promising treatment option that is safe, effective, and unlikely to elicit antiviral resistance. Furthermore, we have preliminary data that suggest it may work similarly during other respiratory virus infections including COVID19/SARS-CoV-2.

In a Phase III Placebo Controlled Clinical Trial with Idiopathic Pulmonary Fibrosis Patients, inhaled sodium pyruvate, a Non-Steroidal Nasal Spray (N115) demonstrated a statistically and clinically significant increase in FEV-1, SaO2, FVC, FEV-1/FVC ratios (from 52% to 86%), and a statistically and clinically significant reduction in coughing, hypoxemia and a reduction in nasal and lung inflammation. Inhaled sodium pyruvate alleviated the symptoms associated with the COVID-19 infections in Patients with COPD and Pulmonary Fibrosis. Nasal Nitric Oxide reduces the rate, duration and severity of viral infections in healthy young children and in healthy adults from the Flu, Rhinovirus and Coronavirus. The literature has reported that Nitric Oxide is elicited and inhibits viral replication in pigs infected with porcine respiratory coronavirus. Additionally Nasal Nitric Oxide levels decreases from normal levels found in healthy adults, in patients with asthma (87%), COPD (73%) CF (44%) and Primary Ciliary Dyskinesia (7%). The rate of infections increases with decreasing levels of nasal nitric oxide. Young children, 6-17 years of age, produce (142%) more nitric oxide than healthy adults, which may explain their resistance to COVID-19. Recently, researchers announced that a high percentage of COVID-19 infected patients that were hospitalized were Diabetics or were Pre-Diabetic. The literature has reported that elevated levels of glucose in patients with diabetes mellitus cause a deficiency in the production of nitric oxide by blunting nitric oxide synthesis, which may explain their susceptibility to COVID-19. Sodium pyruvate increases nitric oxide and is safe for use by Patients with Diabetes. The inhalation of nasal sodium pyruvate increased the synthesis of nasal nitric oxide to normal levels in patients with low levels of nitric oxide to increase all lung functions and decrease the rate of infections.

A clinical survey of 367 patients who took a nasal spray similar to EmphyCorp' s N115 formula, over a two-year period demonstrated a statistically significant decrease in the number, symptoms, and severity of seasonal flu respiratory tract infections. The number of flu or colds was reduced by 70% in Children and approximately 52% in Pregnant Women, Patients with Allergic Rhinitis, Diabetes, and Pulmonary Fibrosis. It has been used successfully by over 3.5 million patients globally in over 200 hospitals during the past 8 years to treat nasal and lung inflammation, congestion in Patients with COPD, Allergic Rhinitis, Pulmonary Fibrosis, sinusitis, the flu and Cystic Fibrosis, with no adverse events reported. It has been used by Children, Diabetics, and Hypertensives, with efficacy and with no known side effects. It has even been shown to be safe for use by Pregnant Women, for whom steroids are contraindicated as they increase the risk of low birth-weight babies.

There are approximately 12 million Americans with COVID-19 Long Hauler Symptoms, including athletes. The symptoms include hypoxemia (low SaO2), fatigue, coughing/sneezing, dyspnea, trouble breathing, body aches, headaches. This chronic disease is referred to as COVID-19 Long Haulers. 7-10% of COVID-19 long haulers are also at serious risk of developing Pulmonary Fibrosis. Conversely, patients with Pulmonary Fibrosis have an increased risk and susceptibility to COVID-19 infection, which can reach a mortality rate of 50%. In a Phase III Clinical Trial in patients in Pulmonary Fibrosis and Idiopathic pulmonary fibrosis, the inhalation of the sodium pyruvate nasal spray demonstrated a statistically and clinically significant improvement in all lung functions, compared to baseline, including an increase in FEV-1, SaO2, FVC, FEV-1/FVC ratios (from 52% to 86%) and a reduction in coughing and fatigue. EmphyCorp/Cellular Sciences Inc. has submitted over 17 human clinicals (Phase I, II, III including animal safety data) to the FDA, demonstrating that the inhalation of sodium pyruvate, significantly reduced respiratory and nasal Inflammation, including oxygen radicals and inflammatory cytokines including IL-6, that causes the so-called cytokine storm COVID-19 patients. Thousands of patients treated with inhaled sodium pyruvate including patients with COPD, Pulmonary Fibrosis, CF, Allergic Rhinitis, Chronic Rhinitis, Sinusitis, and Flu, demonstrated statistically and clinically significant improvement in lung functions with no adverse events reported. This study will examine the effects of N115 (Sodium pyruvate nasal spray) treatment on the symptoms associated with COVID-19 Long Haulers.

ELIGIBILITY:
Inclusion Criteria:

* A prior confirmed positive test for COVID19 and lingering symptoms are required for inclusion.

As outlined on the CDC website, lingering symptoms include:

* Tiredness or fatigue
* Difficulty thinking or concentrating (sometimes referred to as "brain fog")
* Headache
* Loss of smell or taste
* Dizziness on standing
* Fast-beating or pounding heart (also known as heart palpitations)
* Chest pain
* Difficulty breathing or shortness of breath
* Cough
* Joint or muscle pain
* Depression or anxiety
* Fever
* Symptoms that get worse after physical or mental activities

Exclusion Criteria:

* Viral infections other than COVID-19.
* Clinically significant cardiac disease including uncontrolled congestive heart failure and unstable angina
* Pregnancy
* Females of childbearing potential age not on adequate contraception or lactating
* Subjects receiving systemic corticosteroid treatment within one month of Screening Visit
* Subjects Less than 18 years of age
* Hospitalization within last 6 months due to acute exacerbation of airway disease
* Subjects with a clinically significant abnormal chest x-ray within past 12 months
* Medication changes within one month of study entry
* Subjects who have participated in another investigation drug treatment study within the previous month.
* Subjects with a current history of alcohol or recreational drug abuse.
* Subjects who have taken dietary supplements containing pyruvate within 24 hours prior to the screening visit.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Amen, PhD, Study Director — VP of Regulatory Affairs
Locations (1):
- Missouri State University, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abusalamah H, Reel JM, Lupfer CR. Pyruvate affects inflammatory responses of macrophages during influenza A virus infection. Virus Res. 2020 Sep;286:198088. doi: 10.1016/j.virusres.2020.198088. Epub 2020 Jul 4. PMID 32634445
- See also: Summary of previous clinical trials for sodium pyruvate — http://emphycorp.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 patients were enrolled and served as their own baseline control for 7 days followed by 7 days of treatment.
Groups:
- No Treatment First Then Sodium Pyruvate Nasal Spray: All subjects were provided a log for monitoring baseline symptoms associated with Long COVID and asked to record symptom severity using a Likert scale (1-10 with 10 being the most severe) for one week with no treatment. Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 1 and 7 and body temperature recorded twice daily from day 1 to day 7. After recording baseline signs and symptoms for one week without any treatment, all subjects then used N115 20mM sodium pyruvate nasal spray 3x daily for an additional week (day 7-14) and continue to log their symptoms. Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 7 after the first treatment and on day 14. Body temperature continued to be recorded twice daily from day 7 to day 14.
Period: Baseline Day 1-7
Arm/Group | No Treatment First Then Sodium Pyruvate Nasal Spray
Started | 22
Completed | 22
Not Completed | 0
Period: N115 Treatment Day 8-14
Arm/Group | No Treatment First Then Sodium Pyruvate Nasal Spray
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment of COVID19 Long Haulers With Sodium Pyruvate Nasal Spray: This is a single arm, two phased, open label study. All subjects will be provided a log for monitoring baseline symptoms associated with Long COVID and asked to record symptom severity using a Likert scale for one week with no treatment. Vital signs (Blood pressure, temperature, Pulse and SaO2) will be recorded on day 1 and 7. After recording baseline symptoms for one week without any treatment, all subjects will then use N115 20mM sodium pyruvate nasal spray 3x daily for an additional week and continue to log their symptoms. Vital signs (Blood pressure, temperature, Pulse and SaO2) will be recorded on day 7 after the first treatment and on day 14.
Arm/Group | Treatment of COVID19 Long Haulers With Sodium Pyruvate Nasal Spray
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.68 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in the Symptoms of Long COVID-19 Patients
Description: A patient log was used to measure body ache, headache, chills, coughing/sneezing, sore throat, congestion, trouble breathing and other (patient supplied). The patients used a Likert scale from 0 to 10 to assess symptoms with 10 representing the most severe symptom and zero no symptom. The score for each individual symptom was combined into one overall symptom score for the 7 days of baseline (days 1-7) and a separate score for the 7 days of treatment (days 8-14). Therefore, a maximum 7-day score was 70 and a minimum of 0 was possible.
Time Frame: 14 days
Population: Patient scores for baseline days 1-7 of the study when the patients received no treatment were summed into one baseline score (range 0-70). Patient scores for day 8-14 of the study when the patients received 3x daily treatment with 20mM sodium pyruvate were summed into a second score (range 0-70). A Mann-Whitney test was then used to assess statistical difference between baseline and treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray: After recording baseline symptoms for one week (days 1-7) without any treatment, all subjects will then use N115 20mM sodium pyruvate nasal spray 3x daily for an additional week (days 8-14) and continue to log their symptoms. Vital signs (Blood pressure, temperature, Pulse and SaO2) were recorded on day 8 after the first treatment and on day 14.
- Long COVID-19, No Treatment (Baseline): All subjects were provided a log for monitoring baseline symptoms associated with Long COVID and asked to record symptom severity using a Likert scale (0-10 with 10 being the most severe) for one week with no treatment (day 1-7). Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 1 and day 8 prior to treatment and body temperature recorded twice daily from day 1 to day 7.
Arm/Group | Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray | Long COVID-19, No Treatment (Baseline)
Number analyzed (Participants) | 22 | 22
units on a scale
  Body Aches: number analyzed (Participants) | 3 | 3
  Body Aches | 20.33 (4.933) | 27 (5.568)
  Headaches: number analyzed (Participants) | 7 | 7
  Headaches | 15.71 (4.030) | 22.43 (5.062)
  Coughing/Sneezing: number analyzed (Participants) | 11 | 11
  Coughing/Sneezing | 16.09 (8.043) | 28.36 (11.59)
  Sore Throat: number analyzed (Participants) | 1 | 1
  Sore Throat | 9 (0) | 3 (0)
  Trouble Breathing: number analyzed (Participants) | 16 | 16
  Trouble Breathing | 11.88 (7.191) | 27.75 (13.05)
  Congestion: number analyzed (Participants) | 4 | 4
  Congestion | 14.75 (9.032) | 28.25 (19.28)
  Fatigue: number analyzed (Participants) | 3 | 3
  Fatigue | 20.67 (2.517) | 33 (10.82)
  Loss of Smell/Taste: number analyzed (Participants) | 4 | 4
  Loss of Smell/Taste | 23.25 (31.28) | 42 (26.75)
  Anxiety: number analyzed (Participants) | 2 | 2
  Anxiety | 24 (5.657) | 28 (0)
Statistical Analysis 1: Comparison: Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray vs Long COVID-19, No Treatment (Baseline); Body Aches; Test type: Superiority; p = 0.200, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray vs Long COVID-19, No Treatment (Baseline); Headaches; Test type: Superiority; p = 0.0326, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray vs Long COVID-19, No Treatment (Baseline); Coughing/Sneezing; Test type: Superiority; p = 0.0043, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray vs Long COVID-19, No Treatment (Baseline); Trouble Breathing; Test type: Superiority; p = 0.0003, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray vs Long COVID-19, No Treatment (Baseline); Congestion; Test type: Superiority; p = 0.3714, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray vs Long COVID-19, No Treatment (Baseline); Fatigue; Test type: Superiority; p = 0.300, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray vs Long COVID-19, No Treatment (Baseline); Loss of Smell/Taste; Test type: Superiority; p = 0.2286, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray vs Long COVID-19, No Treatment (Baseline); Anxiety; Test type: Superiority; p = 0.999, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Body Temperature in Long COVID-19 Patients
Description: Body temperature will be measured twice daily by thermometer in degrees Fahrenheit. Average body temperature for the first 7 days (days 1-7) was used as a baseline with no treatment and was compared to the average body temperature for the next 7 days (days 8-14) with 20mM sodium pyruvate treatment.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Groups:
- COVID19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray: After recording baseline signs and symptoms for one week without any treatment, all subjects then used N115 20mM sodium pyruvate nasal spray 3x daily for an additional week and continue to log their symptoms. Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 8 after the first treatment and on day 14. Body temperature continued to be recorded twice daily from day 8 to day 14.
- COVID-19 Long Haulers, No Treatment (Baseline): All subjects were provided a log for monitoring baseline symptoms associated with Long COVID and asked to record symptom severity using a Likert scale (0-10 with 10 being the most severe) for one week with no treatment. Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 1 and 8 and body temperature recorded twice daily from day 1 to day 7.
Arm/Group | COVID19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray | COVID-19 Long Haulers, No Treatment (Baseline)
Number analyzed (Participants) | 22 | 22
Degrees Fahrenheit | 98.41 (0.1076) | 98.67 (0.1866)
Statistical Analysis 1: Comparison: COVID19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray vs COVID-19 Long Haulers, No Treatment (Baseline); Test type: Superiority; p < 0.0001, t-test, 2 sided

3. Primary Outcome: Change in Pulse Rate in Long COVID-19 Patients
Description: Patient heart rate will be measured as beats per minute.
Time Frame: Day 1 (1st day Baseline), Day 8 (8th day Baseline), Day 8 (1st day Post-treatment) and Day 14 (7th day post-treatment)
Measure: Mean (Standard Deviation); unit: Beats/minute
Groups:
- COVID19 Long Haulers, Treatment With 20mM Sodium Pyruvate Nasal Spray: After recording baseline symptoms for one week (days 1-7) without any treatment, all subjects will then use N115 20mM sodium pyruvate nasal spray 3x daily for an additional week (days 8-14) and continue to log their symptoms. Vital signs (Blood pressure, Pulse and SaO2) were recorded on day 8 after the first treatment and on day 14. Body temperature was recorded twice daily from day 8-14.
- COVID19 Long Haulers, No Treatment (Baseline): All subjects were provided a log for monitoring baseline symptoms associated with Long COVID and asked to record symptom severity using a Likert scale (0-10 with 10 being the most severe) for one week with no treatment (day 1-7). Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 1 and day 8 prior to treatment and body temperature recorded twice daily from day 1 to day 7.
Arm/Group | COVID19 Long Haulers, Treatment With 20mM Sodium Pyruvate Nasal Spray | COVID19 Long Haulers, No Treatment (Baseline)
Number analyzed (Participants) | 22 | 22
Beats/minute
  Initial reading (day 1 baseline and day 8 treatment) | 80.38 (1.499) | 81.10 (3.463)
  Second reading (day 8 baseline and day 14 treatment) | 79.90 (1.841) | 81.14 (2.330)
Statistical Analysis 1: Comparison: COVID19 Long Haulers, Treatment With 20mM Sodium Pyruvate Nasal Spray vs COVID19 Long Haulers, No Treatment (Baseline); Test type: Superiority; p = 0.1963, ANOVA

4. Primary Outcome: Change in Blood Oxygenation in Long COVID-19 Patients
Description: Blood oxygenation will be measured as %O2 saturation.
Time Frame: Day 1 (1st day Baseline), Day 8 (8th day Baseline), Day 8 (1st day Post-treatment) and Day 14 (7th day post-treatment)
Measure: Mean (Standard Deviation); unit: % Blood oxygen saturation
Groups:
- COVID-19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray: After recording baseline signs and symptoms for one week without any treatment, all subjects then used N115 20mM sodium pyruvate nasal spray 3x daily for an additional week and continue to log their symptoms. Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 7 after the first treatment and on day 14. Body temperature continued to be recorded twice daily from day 8 to day 14.
- COVID-19 Long Haulers, No Treatment (Baseline): All subjects were provided a log for monitoring baseline symptoms associated with Long COVID and asked to record symptom severity using a Likert scale (1-10 with 10 being the most severe) for one week with no treatment. Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 1 and 7 and body temperature recorded twice daily from day 1 to day 7.
Arm/Group | COVID-19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray | COVID-19 Long Haulers, No Treatment (Baseline)
Number analyzed (Participants) | 22 | 22
% Blood oxygen saturation
  Initial reading (day 1 baseline and day 8 treatment) | 96.59 (1.098) | 95.95 (0.8985)
  Second reading (day 8 baseline and day 14 treatment) | 97.59 (0.6661) | 96.09 (0.9211)
Statistical Analysis 1: Comparison: COVID-19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray vs COVID-19 Long Haulers, No Treatment (Baseline); Test type: Superiority; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: COVID-19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray vs COVID-19 Long Haulers, No Treatment (Baseline); Day 1 baseline (day 1 of study) vs Day 1 treatment (day 7 of study); Test type: Superiority; p = 0.0008, Tukey's HSD — Tukey's Multiple comparison test (p-value is adjusted for multiple comparisons)
Statistical Analysis 3: Comparison: COVID-19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray vs COVID-19 Long Haulers, No Treatment (Baseline); Day 1 baseline (day 1 of study) vs Day 7 treatment (day 14 of study); Test type: Superiority; p < 0.0001, Tukey's HSD — Tukey's Multiple comparison test (p-value is adjusted for multiple comparisons)
Statistical Analysis 4: Comparison: COVID-19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray vs COVID-19 Long Haulers, No Treatment (Baseline); Day 7 baseline (day 7 of study) vs Day 1 treatment (day 7 of study); Test type: Superiority; p = 0.0114, Tukey's HSD — Tukey's Multiple comparison test (p-value is adjusted for multiple comparisons)
Statistical Analysis 5: Comparison: COVID-19 Long Haulers, Treatment With Sodium Pyruvate Nasal Spray vs COVID-19 Long Haulers, No Treatment (Baseline); Day7 baseline (day 7 of study) vs Day 7 treatment (day 14 of study); Test type: Superiority; p < 0.0001, Tukey's HSD — Tukey's Multiple comparison test (p-value is adjusted for multiple comparisons)

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray: After recording baseline symptoms for one week (days 1-7) without any treatment, all subjects then used N115 20mM sodium pyruvate nasal spray 3x daily for an additional week (days 8-14) and continued to log their symptoms. Vital signs (Blood pressure, temperature, Pulse and SaO2) were recorded on day 7 after the first treatment and on day 14.
- Long COVID-19, No Treatment (Baseline): All subjects were provided a log for monitoring baseline symptoms associated with Long COVID and asked to record symptom severity using a Likert scale (0-10 with 10 being the most severe) for one week with no treatment (day 1-7). Vital signs (Blood pressure, Pulse, and SaO2) were recorded on day 1 and 7 prior to treatment and body temperature recorded twice daily from day 1 to day 7.
Arm/Group | Long COVID-19, Treatment With 20mM Sodium Pyruvate Nasal Spray | Long COVID-19, No Treatment (Baseline)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT04871815/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT04871815/ICF_001.pdf